CLINICAL TRIAL: NCT03454243
Title: A Study of RXDX-106, an Oral Immunomodulatory TYRO3, AXL, and MER (TAM) Tyrosine Kinase Inhibitor, in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Oral Immunomodulatory Tyrosine Kinase Inhibitor in Patients With Locally Advanced or Metastatic Solid Tumors
Acronym: TITAN
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RXDX-106-01
Record Dates: First submitted 2018-02-21; First posted 2018-03-05 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: Solid Tumors; TYRO3; AXL; MER; Receptor tyrosine kinases (RTKs); Checkpoint inhibitors; Melanoma; Non-small cell lung cancer (NSCLC); Squamous cell carcinoma; Hodgkin lymphoma; Urothelial carcinoma; Microsatellite instability-high carcinomas; TAM Inhibitor
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Hodgkin Disease; Carcinoma, Transitional Cell | interventions — RXDX-106

STUDY DESIGN:
Intervention Model Description: Dose escalation, conventional 3+3 scheme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RXDX-106 (Experimental)
  Interventions: Drug: RXDX-106

INTERVENTIONS:
Drug: RXDX-106 — Patients will receive continuous daily oral doses of RXDX-106 in 21 day cycles. To determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D), study drug will be administered in an escalated fashion starting at dose of 10 mg/day and will proceed at the dose levels prespecified by the dose escalation schema. Once daily dosing for RXDX-106 will initially be tested. However, other dosing schedules (eg, every other day, weight based, etc) may be tested based on safety and PK data to optimize drug exposure.

SUMMARY:
This is a first-in-human, open label, multicenter, dose escalation study of RXDX-106 in patients with locally advanced or metastatic solid tumors, who have no available therapy likely to convey clinical benefit.

This study will examine the safety, tolerability, pharmacokinetics (PK), pharmacodynamics and preliminary efficacy of RXDX 106.

DETAILED DESCRIPTION:
The primary objective of Phase 1 is to assess safety and tolerability, determine the recommended phase 2 dose (RP2D) and assess the pharmacokinetics of RXDX-106. The secondary objective is to evaluate the preliminary antitumor activity of RXDX-106, as assessed by objective response rate (ORR) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and Immune Response Related Criteria in Solid Tumors (iRECIST) in patients with advanced or metastatic solid tumors.

The proposed starting dose of RXDX-106 was calculated based upon nonclinical toxicology studies to determine a recommended first-in-human starting dose, which may be below the biologically active level. Therefore, in order to minimize the number of patients treated at this dose, an accelerated titration design will be used for the first cohort, after which, a conventional 3+3 scheme will be followed for enrollment in subsequent dose levels.

Final determination of the single agent RP2D will be based on available safety, tolerability, PK, pharmacodynamics, and efficacy data from different dose levels and schedules tested, but will be no higher than the maximum tolerated dose. After RP2D has been determined, additional expansion cohorts of patients (up to 15) with specific tumor types, treatment history, and/or expression of a specific biomarker may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumor disease for which standard therapy is not effective, available, acceptable, or is intolerable.
2. Dose level 2 (20 mg) and higher: willing to provide baseline and on treatment tumor biopsies (3 weeks after RXDX-106 treatment initiation), provided the procedure is clinically feasible and not deemed unsafe by the investigator.
3. Prior anticancer therapy is allowed, including prior checkpoint inhibitor treatment.
4. Must have measurable disease per RECIST 1.1 as assessed by computed tomography (CT) scan or magnetic resonance imaging (MRI).

   a. Lesion/s deemed accessible to biopsy for both before and on-treatment biopsies.
5. Males or females aged ≥18 years at screening.
6. Screening laboratory values:

   1. Hemoglobin ≥9 g/dL
   2. Absolute neutrophil count ≥1500 cells/mm3
   3. Platelet count ≥100,000 cells/mm3
   4. Total bilirubin ≤1.5 × upper limit of normal (ULN)
   5. Aspartate aminotransferase and alanine aminotransferase ≤2.5 × ULN
   6. Serum creatinine ≤1.5 mg/dL or estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m2
   7. International Normalized Ratio (INR) or prothrombin time (PT) ≤1.5 × ULN (unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
   8. Activated partial thromboplastin time (aPTT) ≤1.5 × ULN (unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
   9. TSH within normal limits at baseline, (if not WLN, then total T3 or free T3 and free T4 should be within normal limits) or stable with treatment.
7. Patients with treated stable CNS metastases that are asymptomatic (including leptomeningeal carcinomatosis) are allowed, if there is no evidence of progression for at least 4 weeks after CNS-directed treatment as ascertained by clinical examination and brain imaging. Patients requiring steroids must be at a stable or decreasing dose (≤10 mg/day dexamethasone or equivalent) for at least 2 weeks prior to the start of treatment. The use of seizure prophylaxis is allowed.
8. Resolution of any clinically significant toxic effects of prior therapy to grade 0 or 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03 (exception of alopecia and grade 2 peripheral neuropathy).
9. Eastern Cooperative Oncology Group (ECOG) performance status of <2.
10. Other inclusion criteria apply.

Exclusion Criteria:

1. Treated with systemic anticancer therapy or an investigational agent within 2 weeks or 5 half-lives, whichever is shorter, prior to start of study drug treatment. Washout will be 2 weeks for antibody therapy and immunotherapy.
2. Major surgery 21 days or less prior to starting study drug or has not recovered from adverse effects from such procedure.
3. Radiotherapy within 2 weeks prior to start of study drug treatment (palliative radiation or stereotactic radiosurgery within 7 days prior to start of study treatment). Patients must have recovered from all radiotherapy-related toxicities.
4. Has received a live-virus vaccination within 30 days prior to start of study drug treatment.

   a. Seasonal flu and other inactivated vaccines that do not contain live virus are permitted.
5. Severe or unstable medical condition, such as congestive heart failure (New York Heart Association [NYHA] Class III or IV), ischemic heart disease, uncontrolled hypertension, uncontrolled diabetes mellitus, psychiatric condition, as well as an uncontrolled cardiac arrhythmia requiring medication (≥grade 2, according to NCI CTCAE v4.03), myocardial infarction within 6 months prior to starting study treatment, or any other significant or unstable concurrent medical illness that in the opinion of the investigator would preclude protocol therapy.
6. History of non-pharmacologically induced prolonged QTc interval >480 milliseconds.
7. History of other previous or concurrent cancer that would interfere with the determination of safety or efficacy assessment of RXDX-106 with respect to the qualifying solid tumor malignancy.
8. Major active infection requiring parenteral antibiotics.
9. Known HIV infection or active infection with hepatitis B or C. Patients with unknown status at the time of enrollment must be tested during screening.
10. Unable to swallow oral medication.
11. Active gastrointestinal disease (eg, Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would reasonably impact drug absorption.
12. Active autoimmune disease requiring immunosuppressive treatment or history of autoimmune disease requiring immunosuppressive therapy (e.g. requirement for systemic therapy with >10 mg/day prednisone-equivalent) or any other concurrent use of immunosuppressive therapy.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
14. Active retinal pigment epithelium (RPE)/photoreceptor disorders such as; retinitis pigmentosa, cone-rod dystrophies, Bests dystrophy, Stargardt disease (STGD), macular degeneration.
15. Current participation in another clinical study of an investigational agent, vaccine, or device. Concomitant participation in observational studies is acceptable after sponsor approval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Dose Limint Toxicities (DLT) | 21 days following first dose of RXDX-106
  Determine dose-limiting toxicities of RXDX-106
Maximum Tolerated Dose (MTD) | 21 days following first dose of RXDX-106
  Determine MTD of RXDX-106
Recommended Phase 2 Dose (RP2D) | Approximately 12 months
  Determine RP2D of RXDX-106

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 2 years
  Radiographic measurement per RECIST v1.1 and iRECIST as assessed by Investigator
Duration of Response | Approximately 2 years
  Per RECIST v1.1 and iRECIST as assessed by Investigator
Overall Survival (OS) | Approximately 2 years
Progression-Free Survival (PFS) | Approximately 2 years
Maximum observed plasma concentration (Cmax) | Approximately 2 years
Time of maximum observed plasma concentration (Tmax) | Approximately 2 years
AUC throughout dosing interval (AUCτ) | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pratik S. Multani, MD, MS, Study Chair — Chief Medical Officer, Ignyta, Inc.; Sandra Pierina D'Angelo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- START, San Antonio, Texas, United States